CLINICAL TRIAL: NCT02862886
Title: Study of the Effect of Beta-3 Adrenergic Receptor Agonists on Oxidative Stress and Signalling Pathways Implicated in Remodelling of the Uteroplacental Space: Experimental in Vitro Approach on Myometrial Tissue Explants
Acronym: STRESSOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LIONNAIS-COUVREUR AOI 2009
Record Dates: First submitted 2016-08-05; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2011-05

CONDITIONS: Pregnancy

ARMS (1):
- N°1 (Other)
  Interventions: Other: myometrium biopsy

INTERVENTIONS:
Other: myometrium biopsy

SUMMARY:
CHRONOLOGICAL DESCRIPTION OF THE STUDY

1. Information provided to study participants
2. Collection of written informed consent
3. Harvesting of myometrial biopsies
4. Creation of tissue explants using myometrial biopsies
5. Stimulation of the explants with LPS
6. Study of the effect of SAR150640 (beta3-adrenergic agonist) on LPS-induced oxidative stress Moreover, demonstrating the ability of beta3-adrenergic receptor agonists to prevent the appearance of oxidative stress and its consequences on tissues, as a complement to previous studies, is an additional argument for the clinical development of this class of pharmaceuticals in the management of threatened premature delivery and labour induction.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with national health insurance cover
* Patients with a normal pregnancy requiring a caesarean section for obstetrical reasons
* No obvious infectious context

Exclusion Criteria:

* Obvious inflammatory or autoimmune diseases
* Suspected or confirmed infectious context, including HIV, HCV HBV
* Coagulation disorders
* Preexisting or gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
simultaneous assays of 4-amino-5-methylamino-2,7-difluorescein (DAF) / Dihydroethidium (DHE) markers by the technique of high pressure liquid chromatography | The biopsy of myometrium is done specifically for this study in a surgical unit after delivery of the child, in women with a normal pregnancy but requiring a caesarean
  In vitro measurement of the ability of SAR150640 to prevent the release of free radicals (oxidative stress) induced by an inflammatory stimulus on tissue explants of the human myometrium. The level of oxidative stress will be determined using simultaneous assays of DAF/DHE using HPLC. This reference technique for the overall evaluation of oxidative stress is perfectly mastered at the LPPCE (Laboratoire de Physiopathologie et Pharmacologie Cardiovasculaire et Experimentales)

SECONDARY OUTCOMES:
Characterization of signalling pathways induced by oxidative stress during inflammation | The biopsy of myometrium is done specifically for this study in a surgical unit after delivery of the child, in women with a normal pregnancy but requiring a caesarean
  Characterization of the implication of NADPH oxidase (luminometry) and the subunits of NADPH oxidase (gp91, p22fox, p67phox, p47phox, p40phox as well as Rac1/2) and NO synthases (eNOS & iNOS), as the source of the oxidative stress induced by an inflammatory stimulus, using Western blot

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France